CLINICAL TRIAL: NCT01930552
Title: A Phase I Study of the Safety, Tolerability, and Pharmacokinetics of Aflibercept in Combination With FOLFIRI Administrated Every 2 Weeks in Chinese Patients With Advanced Solid Malignancies
Brief Title: A Phase I Study of Aflibercept Plus FOLFIRI (Irinotecan, 5-Fluorouracil, and Leucovorin) in Chinese Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD11470; U1111-1115-7286 (Other: UTN)
Record Dates: First submitted 2013-08-14; First posted 2013-08-29 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms | interventions — aflibercept; Leucovorin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort 1 (Experimental): aflibercept IV infusion for 1 hour followed by FOLFIRI IV infusion every 2 weeks
  Interventions: Drug: Aflibercept AVE0005; Drug: Leucovorin; Drug: Irinotecan; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: Aflibercept AVE0005 — Pharmaceutical form:Solution for infusion Route of administration: Intravenous
Drug: Leucovorin — Pharmaceutical form:Solution for infusion Route of administration: Intravenous
Drug: Irinotecan — Pharmaceutical form:Solution for infusion Route of administration: Intravenous
Drug: 5-Fluorouracil — Pharmaceutical form:Solution for infusion Route of administration: Intravenous

SUMMARY:
Primary Objective:

To assess the safety and pharmacokinetics preliminarily of the dose of intravenous (IV) aflibercept used in western studies in combination with FOLFIRI (Irinotecan, 5-Fluorouracil, and Leucovorin) given intravenously every 2 weeks in Chinese patients with solid tumors.

Secondary Objectives:

* To make a preliminary assessment of antitumor effects of the combination of FOLFIRI plus aflibercept in patients with measurable disease (RECIST 1.1).
* To evaluate the immunogenicity of IV aflibercept.

DETAILED DESCRIPTION:
Total duration of the study per patient is in the range of 17 to 29 weeks.

This trial is being conducted in China, where the INN designation for the study molecule is "aflibercept" and this term is therefore used throughout the synopsis. In the US, the US proper name is "ziv-aflibercept".

ELIGIBILITY:
Inclusion criteria:

- Histologically or cytologically confirmed solid malignancy that is metastatic or unresectable for which FOLFIRI (Irinotecan, 5-Fluorouracil, and Leucovorin) treatment is appropriate

Exclusion criteria:

* Treatment with chemotherapy, hormonal therapy, radiotherapy, surgery, or an investigational agent within 28 days
* Eastern Cooperative Oncology Group (ECOG) >1
* Need for a major surgical procedure or radiation therapy during the study
* Diagnosis of squamous-cell lung cancer
* Cumulative radiation therapy to > 25% of the total bone marrow
* History of brain metastases
* Inadequate organ and bone marrow function
* Uncontrolled hypertension
* Evidence of clinically significant bleeding diathesis or underlying coagulopathy
* Prior FOLFIRI treatment but have not been appropriate for safety reasons
* Patients with known Gilbert's syndrome

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with standard safety assessments (adverse events and laboratory tests) | Up to last treatment + 30 days
Pharmacokinetics: Assessment of plasma concentrations of aflibercept, CPT-11 (irinotecan) and Fluorouracil (5-FU) | Up to last aflibercept administration + 90 days

SECONDARY OUTCOMES:
Anti-tumor activity assessment - overall response rate | Up to 17 Weeks
Anti-tumor activity assessment - duration response | Up to 17 Weeks
Anti-aflibercept antibody detection | Up to last aflibercept administration + 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- China (2):
  - Investigational Site Number 156002, Beijing
  - Investigational Site Number 156001, Guangzhou